CLINICAL TRIAL: NCT00775736
Title: Observational Study Evaluating Safety in Patients With Type 2 Diabetes Treated With NovoMix® 30 or NovoMix® 50 or NovoMix®70 (Biphasic Insulin Aspart)
Brief Title: Observational Study Evaluating the Safety of NovoMix® in Type 2 Diabetes Patients Previously Treated With a Human Premix Insulin
Acronym: Mix2Mix
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-3665
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 50; Drug: biphasic insulin aspart 70

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Start dose and frequency and safety data collection at the discretion of the physician following clinical practice
  Other Names: BIAsp
Drug: biphasic insulin aspart 50 — Start dose and frequency and safety data collection at the discretion of the physician following clinical practice
Drug: biphasic insulin aspart 70 — Start dose and frequency and safety data collection at the discretion of the physician following clinical practice

SUMMARY:
This study is conducted in Europe. The objective of this observational study is to evaluate the number of serious side effects, when initiating NovoMix® treatment in patients with type 2 diabetes who previously used a human premix insulin under normal clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus

Exclusion Criteria:

* Known or suspected allergy to study product or related products.
* Pregnancy or breastfeeding or intention of becoming pregnant within the next 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: After the participating physicians' decision has been made to initiate NovoMix® therapy, any patient with type 2 diabetes who is currently treated with a human premix insulin therapy.
Sampling Method: Non-Probability Sample
Enrollment: 611 (Actual)
Dates: Start 2008-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The number of serious adverse drug reactions, including major hypoglycaemic episodes, reported during the study period. | At baseline, 12 and 26 weeks.

SECONDARY OUTCOMES:
Number of all hypoglycaemic episodes. | At baseline, 12 and 26 weeks.
Number of all adverse drug reactions. | At baseline, 12 and 26 weeks.
HbA1c | at 12 and 26 weeks
Evaluation of fasting plasma glucose (FPG) values and postprandial glucose (PPG) levels | at 12 and 26 weeks
Weight changes | at 12 and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Novo Nordisk Investigational Site, Brussels, Belgium
- Novo Nordisk Investigational Site, Luxembourg, Luxembourg

REFERENCES:
- [Result] Nobels F, D'Hooge D, Crenier L. Switching to biphasic insulin aspart 30/50/70 from biphasic human insulin 30/50 in patients with type 2 diabetes in normal clinical practice: observational study results. Curr Med Res Opin. 2012 Jun;28(6):1017-26. doi: 10.1185/03007995.2012.695730. Epub 2012 Jun 11. PMID 22612579
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com